CLINICAL TRIAL: NCT00054444
Title: A PHASE I STUDY OF PELVIC RADIATION THERAPY WITH CONCOMITANT WEEKLY CISPLATIN AND TOPOTECAN CHEMOTHERAPY IN PATIENTS WITH CERVICAL CARCINOMA WITHOUT EXTRA-PELVIC METASTASIS
Brief Title: Radiation Therapy and Chemotherapy in Treating Patients With Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9913; NCI-2009-00617 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000270680; GOG-9913; GOG-9913 (Other: Gynecologic Oncology Group); GOG-9913 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Squamous Cell Carcinoma; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Conformal; Cisplatin

ARMS (1):
- Treatment (topotecan hydrochloride, radiation, cisplatin) (Experimental): Patients undergo radiotherapy 5 days a week for 6 weeks. Patients receive cisplatin IV and topotecan IV over 30 minutes once weekly for a total of 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Topotecan Hydrochloride Liposomes; Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Topotecan Hydrochloride Liposomes — Given IV
  Other Names: Brakiva
Radiation: 3-Dimensional Conformal Radiation Therapy
  Other Names: 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Cisplatin — Given IV

SUMMARY:
This phase I trial is studying the side effects and best way to give radiation therapy when given together with topotecan and cisplatin in treating patients with locally advanced cervical cancer. This trial is also studying the best dose of topotecan when given in this regimen. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as topotecan and cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of pelvic radiotherapy, cisplatin, and topotecan in patients with locally advanced cervical cancer.

II. Determine the maximum tolerated dose (MTD) of topotecan when administered in this regimen in this patient population.

SECONDARY OBJECTIVES:

I. Determine the site of recurrence (local vs distant) in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of topotecan.

Patients undergo radiotherapy 5 days a week for 6 weeks. Patients receive cisplatin IV and topotecan IV over 30 minutes once weekly for a total of 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 6 patients experiences dose-limiting toxicity. Once the MTD is determined, an additional cohort of 20 patients receives treatment as above at the MTD.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary invasive carcinoma of the uterine cervix

  * Stages IB2, II, IIIB, and IVA disease
  * Any cell type
* No known metastasis to scalene nodes or organs outside the radiation field
* No known intraperitoneal metastases
* No evidence of extrapelvic disease based on negative CT or PET scan
* Must enroll within 8 weeks of diagnosis
* Performance status - GOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine normal
* Creatinine clearance > 50 mL/min
* Prior ureteral obstruction allowed provided stent or nephrostomy tube has been placed
* No renal abnormalities, such as pelvic kidney, horseshoe kidney, or prior renal transplantation that would require modification of radiation fields
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No septicemia or severe infection
* No other medical or psychiatric condition that would preclude study compliance
* No prior chemotherapy for any prior malignancy
* No prior cytotoxic chemotherapy for this malignancy
* No prior radiotherapy for any prior malignancy
* No prior pelvic or abdominal radiotherapy for this malignancy
* No prior therapy for this malignancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with acute toxicity assessed by Common Terminology Criteria for Adverse Events version 3.0 | Up to 30 days after completion of radiation therapy
Incidence of patients with chronic toxicity assessed by Common Toxicity Criteria Radiation Therapy Oncology Group/European Organisation for Research and Treatment of Cancer (CTC RTOG/EORTC) | Up to 5 years

SECONDARY OUTCOMES:
Site of treatment failure | Up to 5 years
  Identified as local versus distant.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rose, Principal Investigator — Gynecologic Oncology Group
Locations (10):
- United States (10):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma